CLINICAL TRIAL: NCT06556459
Title: Psychological and Psychopathological Characteristics of Patients With Severe or Pathological Obesity Candidates for Bariatric Surgery
Brief Title: Psychological and Psychopathological Characteristics of Patients With Obesity Candidates for Bariatric Surgery
Acronym: PSICOBAR
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6678
Record Dates: First submitted 2024-07-26; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric Surgery — The patient performs:
  * psychological clinical interview
  * psychodiagnostic examination
  * internal medical examination
  * blood tests
  * electrocardiogram
  * bariatric surgery
  * surgical visit

SUMMARY:
Patients with obesity who are candidates for bariatric surgery may exhibit high rates of psychological symptoms, mostly anxiety and depression, and even full-blown mental disorders. The etiopathogenesis of this association has been variously investigated, and among the various factors, the presence of systemic inflammation, even if low-grade, seems to be an underlying mechanism for both conditions. These associations have been shown to have a significant impact from both a clinical perspective and regarding the outcomes of the surgery itself . Worse outcomes have been described in individuals with anxiety-depressive syndromes or mood disorders. However, additional impacts on treatment can also result from the presence of dysfunctional personality traits and early traumatic experiences (reported in about 50% of individuals with severe/pathological obesity), which, in turn, correlate with pathological eating behaviors in a high percentage of cases.

Studies conducted in various countries show that about 40% of all patients undergoing bariatric surgery have at least one psychiatric diagnosis, with depressive disorders, anxiety disorders, and eating disorders being the three most common diagnoses

Most studies on bariatric patients have focused on factors predisposing to severe obesity or predictive of surgical outcomes and post-surgery progress, but often lack a more precise psychological and psychopathological characterization of this patient population. Targeted studies with a longitudinal design that include long-term post-surgery follow-up are necessary to clarify the actual role of these factors as well as their interaction with other pathophysiological mechanisms involved in the clinical presentation and response to various treatment strategies. Identifying new therapeutic targets during the preoperative evaluation process could, in fact, contribute to improving clinical and post-surgical outcomes. Despite bariatric surgery demonstrating a positive short-term impact on weight-related comorbidities and functioning levels, particularly in social relationships, the emergence of unique and peculiar psychosocial problems and/or concerns in the postoperative follow-up has been reported. In a 10-year longitudinal study, a significant increase in mental health service access was observed following bariatric surgery, especially among those with a positive psychiatric history before the surgery.

Besides weight loss, surgical outcomes should include improvements in metabolic status and medical comorbidities, increased quality of life, and better psychosocial and behavioral functioning. Even in a patient with excellent postoperative weight loss, psychosocial problems such as disruptions in interpersonal relationships, body image dissatisfaction, substance use, or suicidal ideation may arise.

Therefore, this study aims to investigate the sociodemographic, clinical, personality, psychological, and psychopathological characteristics of patients with severe/pathological obesity requesting bariatric surgery through a baseline assessment and, if applicable, at six and twelve months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* All sex;
* Age ≥18 years
* Diagnosis of grade II or grade III (or pathological) obesity based on body mass index values, respectively, of 35-40 and >40 kg/m²
* Multidisciplinary evaluation aimed at indicating bariatric surgery interventions as per clinical practice
* Provision of written informed consent to participate in the study

Exclusion Criteria:

* Age <18 years
* Diagnosis of neurological disorders associated with cognitive decline (such as to impair the execution of psychometric assessment)
* Confirmed pregnancy, breastfeeding, or potential pregnancy with positive serological β- HCG
* Refusal to sign the informed consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosis of grade II or grade III (or pathological) obesity based on body mass index values, respectively, of 35-40 and >40 kg/m² who access the Policlinico to apply for bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of anxiety and depressive symptoms with Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 Questionnaire (GAD-7), Beck's Depression Inventory (BDI-II) and State-Trait Anxiety Inventory (STAI Y). | 1 year
  Evaluation of changes in anxiety and depressive symptoms from baseline to one year after bariatric surgery with Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 Questionnaire (GAD-7), Beck's Depression Inventory (BDI-II) and State-Trait Anxiety Inventory (STAI Y).
  GAD - 7:
  0 - 4: minimal 5 - 9: mild 10 - 14: moderate 15 - 21: severe
  PHQ - 9:
  0 - 4: minimal 5 - 9: mild 10 - 14: moderate 15 - 19: moderately severe 20 - 27: severe
  BDI-II:
  < 7: none 8 - 17: mild 18 - 24: moderate >25: severe
  STAI-Y1/Y2:
  20 - 37: none or minimal 38 - 44: moderate 45 - 80: severe
Interim evaluation of anxious and depressive symptoms with Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 Questionnaire (GAD-7), Beck's Depression Inventory (BDI-II) and State-Trait Anxiety Inventory (STAI Y). | 6 months
  Interim evaluation of anxiety and depressive symptoms at six months after bariatric surgery with Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder-7 Questionnaire (GAD-7), Beck's Depression Inventory (BDI-II) and State-Trait Anxiety Inventory (STAI Y).
  GAD - 7:
  0 - 4: minimal 5 - 9: mild 10 - 14: moderate 15 - 21: severe
  PHQ - 9:
  0 - 4: minimal 5 - 9: mild 10 - 14: moderate 15 - 19: moderately severe 20 - 27: severe
  BDI-II:
  < 7: none 8 - 17: mild 18 - 24: moderate >25: severe
  STAI-Y1/Y2:
  20 - 37: none or minimal 38 - 44: moderate 45 - 80: severe

SECONDARY OUTCOMES:
Evaluation of changes in psychological and psychopathological state dimensions from baseline to one year after bariatric surgery. | 1 year
  Evaluation of changes in other psychological and psychopathological state dimensions from baseline to one year after bariatric surgery with Short Form Health Survey - 36 (SF-36), Perceived Stress Scale (PSS), Eating Disorder Examination Questionnaire (EDE-Q 6), Binge Eating Scale (BES), Clinical Impairment Assessment Questionnaire (CIA 3.0), Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM).
  SF-36:
  The score ranges from 0 (negative health) to 100 (positive health).
  PSS:
  0-13: low stress 14-26: moderate stress 27-60: high perceived stress
  EDE-Q 6:
  > 2,8: clinically significant
  BES:
  <17: improbable 17-27: possible >27: possible
  CIA 3.0:
  The resulting scores range from 0 to 48, where a higher score indicates a higher level of secondary psychosocial impairment.
  CORE-OM:
  <0,6: healthy 0,6-1: low 1-1,5: mild 1,5-2: moderate 2-2,5: moderately severe >2,5: severe
Interim evaluations of changes in other psychological and psychopathological state dimensions at six months after bariatric surgery. | 6 months
  Interim evaluations after six months of changes in other psychological and psychopathological state dimensions as per clinical practice.
  It will be used Short Form Health Survey - 36 (SF-36), Perceived Stress Scale (PSS), Eating Disorder Examination Questionnaire (EDE-Q 6), Binge Eating Scale (BES), Clinical Impairment Assessment Questionnaire (CIA 3.0), Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM).
  SF-36:
  The score ranges from 0 (negative health) to 100 (positive health).
  PSS:
  0-13: low stress 14-26: moderate stress 27-60: high perceived stress
  EDE-Q 6:
  > 2,8: clinically significant
  BES:
  <17: improbable 17-27: possible >27: possible
  CIA 3.0:
  The resulting scores range from 0 to 48, where a higher score indicates a higher level of secondary psychosocial impairment.
  CORE-OM:
  <0,6: healthy 0,6-1: low 1-1,5: mild 1,5-2: moderate 2-2,5: moderately severe >2,5: severe
Evaluation of the variation in global functioning levels from baseline to six months after bariatric. | 6 months
  Evaluation of the variation in global functioning levels from baseline at six months after bariatric surgery with Difficulties in Emotion Regulation Scale (DERS), Barratt Impulsiveness Scale (BIS 11), Connor-Davidson Resilience Scale (CD-RISC) and Childhood Trauma Questionnaire (CTQ-SF).
  DERS:
  Higher scores suggest greater problems with emotion regulation
  BIS-11:
  30-49: low 50-69: mild 70-89: severe 90-120: extremely severe
  CD-RISC:
  A higher score indicates a higher level of resilience
  CTQ-SF:
  This questionnaire measures five types of abuse. For each type of childhood trauma, the higher the score is, the greater the severity of abuse for that scale.
Evaluation of the variation in global functioning levels at one year after bariatric surgery. | one year
  Evaluation of the variation in global functioning levels from baseline at one year after bariatric surgery with Difficulties in Emotion Regulation Scale (DERS), Barratt Impulsiveness Scale (BIS 11), Connor-Davidson Resilience Scale (CD-RISC) and Childhood Trauma Questionnaire (CTQ-SF).
  DERS:
  Higher scores suggest greater problems with emotion regulation
  BIS-11:
  30-49: low 50-69: mild 70-89: severe 90-120: extremely severe
  CD-RISC:
  A higher score indicates a higher level of resilience
  CTQ-SF:
  This questionnaire measures five types of abuse. For each type of childhood trauma, the higher the score is, the greater the severity of abuse for that scale.
Evaluation of the variation of the quality of life at six months after bariatric surgery with Short Form Health Survey - 36 (SF-36). | six months
  Evaluation of the variation of the quality of life at six months after bariatric surgery with Short Form Health Survey - 36 (SF-36).
  SF-36:
  The score ranges from 0 (negative health) to 100 (positive health).
Evaluation of the variation of the quality from baseline to one year after bariatric surgery with Short Form Health Survey - 36 (SF-36). | 1 year
  Evaluation of the variation of the quality from baseline to one year after bariatric surgery with Short Form Health Survey - 36 (SF-36).
  SF-36:
  The score ranges from 0 (negative health) to 100 (positive health).
Identification of correlation between psychological and psychopathological trait dimensions and metabolic and inflammatory correlates. | 1 year
  Identification of correlation between psychological and psychopathological trait dimensions and metabolic and inflammatory correlates that predict response to bariatric surgery interventions.
  It will be measured the variation of the metabolic and inflammatory correlates from baseline to one year after bariatric surgery.
  It will be considered: complete blood count with leukocyte count; C-reactive Protein (PCR); Erythrocyte sedimentation rate (VES); fibrinogen; magnesium; calcium; phosphorus; parathyroid hormone (PTH); vitamin D; uric acid; carbohydrate and lipid profile (glucose, total and HDL cholesterol, triglycerides);

CONTACTS AND LOCATIONS:
Overall Officials: Marco Raffaelli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Chirurgia Endocrina e Metabolica, Roma, Italy